CLINICAL TRIAL: NCT00220402
Title: Long-Term Open-Label Extension Trial for Subjects Completing the Phase 3 Trial of Fesoterodine (SP583) for the Treatment of Overactive Bladder Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: SP738
Record Dates: First submitted 2005-08-30; First posted 2005-09-22 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Overactive Bladder Syndrome

INTERVENTIONS:
Drug: SPM 907

SUMMARY:
This trial will provide long-term data on safety, satisfaction and maintenance on therapy of fesoterodine (SPM 907) in subjects with overactive bladder syndrome.

Subjects completing the 12 week treatment period of SP583 had the opportunity to participate if eligibility was confirmed. They received fesoterodine 8mg with the option to reduce the dose to 4mg during scheduled visits, and to increase again to 8mg, a procedure which could be followed on an annual basis.

Two primary efficacy variables will be assessed, which are observation and assessment of adverse events and duration on therapy.

Secondary efficacy parameters included various parameters derived from micturition diaries and the evaluation of Quality of Life questionnaires (KHQ and ICIQ-SF).

The most important safety variables included the assessment of adverse events, laboratory parameters, changes in ECG, physical exams and measurement of residual urine.

ELIGIBILITY:
Inclusion Criteria:

* Participated in SP583

Exclusion Criteria:

* Failure to complete 12 week treatment with SPM 907

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Steinert, Study Director — UCB Pharma
Locations (1):
- Schwarz, Monheim, Germany